CLINICAL TRIAL: NCT06489977
Title: Rigid Corset Immobilisation of Patients Suffering From Spondylodiscitis: Practice Assessment
Acronym: Cors'aime
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: M24RC0512
Record Dates: First submitted 2024-06-24; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Management of Spondylodiscitis
Keywords: spondylodiscitis; corset; spinal infection; vertebral disc; spinal bodies; practical assessment
MeSH Terms: conditions — Discitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study is a survey of the current management of patients suffering from spondylodiscitis.

DETAILED DESCRIPTION:
Our main objective was to describe the use of rigid corsets to immobilise patients with spondylodiscitis in hospital, by asking doctors about their practices.

The secondary objectives are :

* To describe the use of rigid corsets to immobilise patients suffering from spondylodiscitis in hospital by asking paramedical staff about the way in which medical prescriptions were implemented and patients about their compliance.
* To measure the rate of satisfaction and understanding of patients treated with a corset.
* To detail the different ways in which doctors and paramedical staff manage patients hospitalised for spondylodiscitis, depending on their age, training, speciality and the department in which they work.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Patients aged over 18,
* Patients hospitalised at Clermont-Ferrand University Hospital with infectious spondylodiscitis,
* Patient willing to be interviewed.

For care workers:

- Doctors, nurses or care assistants involved in the care of patients hospitalised with spondylodiscitis.

Exclusion Criteria:

For patients :

* Minor patients,
* Patients wearing a corset for a non-infectious spinal pathology,
* Patient refusing to take part in the study.

For care workers:

- Doctor, nurse or nursing auxiliary refusing to take part in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Medical and paramedical staff working in facilities providing care for patients hospitalised with spondylodiscitis will be asked to complete a questionnaire assessing their day-to-day practices.
  Patients who have been hospitalised for spondylodiscitis in the Infectious Diseases and Rheumatology Departments at Clermont-Ferrand University Hospital during the last 4 years will receive the information note. After a period of one month, if they have not expressed their opposition, they will be contacted by telephone to take part in a semi-structured interview lasting 15 to 20 minutes to find out about their experience of care and their satisfaction.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Physician survey to identify medical practices in the management of patients suffering from spondylodiscitis in hospital. | 3 months
  Questionnaire to evaluate medical practices

SECONDARY OUTCOMES:
Practical application of rigid corset prescriptions by paramedical teams. | 3 months
  Questionnaire to evaluate paramedical practices
Patient compliance, feedback, understanding and satisfaction with wearing the corset | 3 months
  Questionnaire to assess patient compliance and feelings

CONTACTS AND LOCATIONS:
Overall Officials: Aurore MIGNE, Principal Investigator — University Hospital, Clermont-Ferrand; Orlane MENAGE, Principal Investigator — University Hospital, Clermont-Ferrand; Clémence RICHAUD, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France